CLINICAL TRIAL: NCT07005089
Title: Diagnostic Accuracy of Ultrasound and Tumors Markers in Diagnosis of Complex Ovarian Cysts in Adolescent, Histopathological Correlation
Brief Title: Diagnostic Accuracy of Ultrasound and Tumors Markers in Diagnosis of Complex Ovarian Cysts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Fathy Ibrahim Mohamed, Resident of Obstetrics and Gynecology, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Complex Ovarian Cysts
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2023-02

CONDITIONS: Complex Ovarian Cyst
MeSH Terms: interventions — Laparotomy; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cases with Complex Ovarian Cyst (Experimental): About 48 female patients suffered from Complex Ovarian Cysts. tumor marker and MRI should be done. If no suspicion of cancer by tumor markers and the patient was Symptomatic and the size of the cysts >5 cm: Laparotomy or Laparoscopic cystectomy and histopathological examination were done.
  Interventions: Procedure: Laparotomy or laparoscopic ovarian cystectomy

INTERVENTIONS:
Procedure: Laparotomy or laparoscopic ovarian cystectomy — to evaluate diagnostic accuracy of ultrasound and tumors markers in diagnosis of complex ovarian cysts in adolescent with histopathological correlation.
  Other Names: ultrasound and tumors markers

SUMMARY:
Cystic ovarian lesions are more common in adolescences due to onset of hormonal activity in prepubertal age. Most cysts are functional but a malignant etiology must nevertheless always be eliminated.

Most ovarian cysts in adolescents are benign in nature, with 60% being simple ovarian cysts.

Cystic neoplasia may be benign, borderline, or malignant. The large majority are benign or borderline, accounting for 80% and 16%, respectively

DETAILED DESCRIPTION:
Cystic ovarian lesions are more common in adolescences due to onset of hormonal activity in prepubertal age. Most cysts are functional but a malignant etiology must nevertheless always be eliminated.

Complex benign cysts are about 16% of all ovarian cysts, :(mature cystic teratoma 55-70%, endometrioma, gonadoblastoma, serous cystadenoma, mucinous cystadenoma, cystadenoﬁbroma).

About 1% of ovarian tumors can be malignant and differential diagnosis with benign ones is sometimes difficult. Concerning the management of such tumors in adolescents for which future fertility is a concern.

Malignant ovarian tumors types are :( Sex cord-stromal tumors:( juvenile granulosa cell tumor is most common about 50% and Sertoli-Leydig cell tumor), Germ cell tumors: (dysgerminoma30%, immature teratoma30%, yolk sac tumor, embryonal carcinoma and polyembryoma) and Epithelial tumors:(serous adenocarcinoma, mucinous adenocarcinoma).

Ultrasonography is a gold standard modality in the evaluation of the female pelvis in adolescence today the method of choice for distinguishing between benign and malignant adnexal pathologies. Using pattern of recognition several types of cysts and tumors can be recognized according to their characteristic appearance.

If a complex ovarian cyst is diagnosed on an ultrasound scan, magnetic resonance imaging (MRI) of the pelvis should be requested. MRI provides good soft tissue delineation and allows identification of the ovarian tumor type, MRI had excellent performance and positive correlation, but significant interobserver variability remains.

The discovery of reliable ovarian cancer biomarkers plays a crucial role in the disease diagnosis, management and strongly impact in patient's prognosis and survival as (lactate dehydrogenase, beta human chorionic gonadotrophin, alpha fetoprotein and ca-125).

Lactate dehydrogenase is widely recognized that the increased rate of glycolysis in rapidly growing tumor as Dysgerminoma and Immature teratoma.

Alpha fetoprotein (AFP) and ß-human chorion gonadotropin (ß-HCG) are markers of tumorous lesions of the ovary. AFP can be a marker of immature ovarian teratoma, yolk sac tumor, and embryonal carcinoma. ß-HCG can be a marker of malignant germ cell tumors, choriocarcinoma, and embryonal cell carcinomas.

CA-125 The most extensively studied ovarian cancer associated marker which detecting Epithelial tumors.

Final diagnoses only by histopathological examination, Ovarian cancer is a very heterogeneous disease and is mainly represented four main distinct histological subtypes: serous, the most frequent; endometrioid; mucinous and clear cells. In some cases, it is present a mixture of these histological types. Each of these histological subtypes may exhibit a different degree of differentiation.

ELIGIBILITY:
Inclusion Criteria:

* Female patients diagnosed by complex ovarian cysts

Exclusion Criteria:

* simple ovarian cyst < 7cm
* Any suspected ovarian malignancy

Ages: 11 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Diagnosis of Complex Ovarian Cysts | 3 months
  Assessment and Diagnosis of female patients with Complex Ovarian Cysts by ultrasound or tumor markers

CONTACTS AND LOCATIONS:
Overall Officials: El kotb Hassan El kotb El saedy, Professor, Study Chair — Al-Azhar Faculty of medicine,Assuit
Locations (1):
- Al-Azhar University hospital, Asyut, Egypt